CLINICAL TRIAL: NCT02932540
Title: The Effects of Head Positioning on Beat to Beat Cerebral Haemodynamics: a Comparison Between Acute Stroke Patients and Healthy Control Subjects
Brief Title: Head Position on Cerebral Haemodynamics in Acute Ischemic Stroke and Controls
Status: Completed | Type: Observational
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0538
Record Dates: First submitted 2016-10-06; First posted 2016-10-13 (Estimated); Last update posted 2020-01-30 (Actual); Status verified 2016-05

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Healthy controls: healthy controls subjects who have age, sex and Blood pressure matched with the acute ischaemic stroke patient
  Interventions: Other: change of head position
- AIS patient-transient arm: transient change of head position from lying flat (0 degree) to sitting up (30 degree)
  Interventions: Other: change of head position
- AIS patient - persistent lying flat: lying flat (0 degree) head position for the first 24 hours in the hospital admission
  Interventions: Other: change of head position
- AIS patient - persistent sitting up: sitting up ( 30 degree) head position for the first 24 hours in the hospital admission
  Interventions: Other: change of head position

INTERVENTIONS:
Other: change of head position — patient can be allocated to the transient change of the head position, persistent lying flat position in the first 24 hours of the hospital admission and persistent sitting up in the first 24 hours of the hospital admission

SUMMARY:
Cerebral autoregulation is an important mechanism whereby cerebral perfusion is normally maintained at a constant level, over a relatively wide blood pressure range. It can be assessed noninvasively by the use of Trans Cranial Doppler (TCD). This means using ultrasound probes over both sides of the head to measure changes in blood flow in one of the main brain arteries (the middle cerebral artery) in response to beat to beat changes in blood pressure dynamic cerebral autoregulation (dCA). It is established that dCA is impaired following moderate to severe stroke, acting as a key role in the development of secondary brain damage related to brain swelling and further damage related to the low blood flow. The administration of clot busting therapy (thrombolysis), one of the main approved treatments of acute ischaemic stroke (AIS), results in recanalisation of the blocked artery in only approximately 50% of patients. Therefore, as well as attempts to treat major vessel blockage, improving brain blood flow, particularly to the penumbral area, through arteries that bypass the blockage is another potential therapeutic approach in AIS.One simple way of achieving this might be to lower the head of AIS patient into a lying flat (0⁰) position. However, to date, there have been very few studies exploring this. This research will use the noninvasive technique of Trans Cranial Doppler (TCD) to see how blood flow changes in different head positions, both in healthy volunteers and AIS patient. This study will provide important data regarding blood pressure management in acute stroke, an important and common clinical dilemma.

DETAILED DESCRIPTION:
In the United Kingdom (UK) alone, approximate 100,000 people suffer a stroke each year. Improved management of stroke patients not only reduces morbidity and mortality, but also reduces the cost of long term social care.

The brain has control systems (i.e.cerebral autoregulation) to maintain blood flow to the brain, over a relatively wide blood pressure range. Cerebral Autoregulation can be described as static, reflecting the integrity of such mechanisms over time, or dynamic, occurring in response to sudden fluctuations in perfusion pressure. When blood pressure drops, small arteries increase in size to restore flow levels, and when blood pressure rises, they narrow to protect the most delicate blood vessels. It is known that sudden decompensated blood pressure (BP) changes can occur after stroke, this could result in brain bleeding and swelling when there is uncontrolled increased blood flow, or reduce the viability of tissue surrounding the stroke area when there is reduced blood flow to the brain.

It is known that the clot busting agent (Alteplase), the main effective treatment used in the acute stroke can only improve blood flow in already blocked arteries in 50% of patients. Therefore, as well as attempts to treat blockage of major vessel, improving the blood flow through vessel that bypass the blocked vessel around the stroke area (penumbra) could be another potential therapeutic approach in acute ischaemic stroke patients. A simple way of increase blood flow to these penumbral area might be just lower the head of acute stroke patients into a lying flat position. Several observational studies have investigated the effects of head positioning on blood flow to the brain in a healthy population, however few studies carried out on acute ischaemic stroke patients so far.

Cerebral autoregulation can be assessed non-invasively by the use of Trans Cranial Doppler (TCD). This means using ultrasound probes over both sides of the head to measure changes in blood flow in one of the main brain arteries (the middle cerebral artery) in response to beat to beat changes in blood pressure dynamic cerebral autoregulation. This research will use the noninvasive technique of Trans Cranial Doppler to see how blood flow changes during different head position between acute ischaemic stroke patients and healthy controls, as well as over time during recovery after a stroke. This knowledge will help us to understand the changes in brain blood flow control and blood pressure in stroke patients, with implications of diagnosis, prognosis, and treatment of the disease.

ELIGIBILITY:
Inclusion Criteria:

- Informed volunteer consent, patient consent or personal consultee declaration form

* Male or female, aged 18 years or above
* Able (in the Investigator's opinion) and willing to comply with all study requirements
* Willing to allow his or her General Practitioner (GP) to be notified of participation in the study Stroke Patient-specific Inclusion Criteria
* Clinical diagnosis of ischaemic stroke within 24 hours of onset (for patients waking with a stroke, time of onset will be taken to be the time when the patient was last asymptomatic)

Exclusion Criteria:

* Male or Female, aged under 18 years

  * Unable (in the Investigator's opinion) or unwilling to comply with any study requirements
  * Participants who practice yoga regularly
  * Female participants who are pregnant, lactating or planning pregnancy during the course of the study Stroke Patient-specific Exclusion Criteria
  * Clinical diagnosis of stroke greater than 24 hours from onset
  * Having had a resolved transient ischaemic attack (TIA) (i.e. neurological symptoms completely resolved upon hospital presentation)
  * Definite clinical indication to 'sitting up' (≥30⁰) head position (i.e. pneumonia, decompensated heart failure)
  * Definite clinical indication to lying flat (0⁰) head position (i.e. shock, airways obstruction)
  * Co-morbidity with anticipated life expectancy less than 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 11 healthy control subjects 11 acute ischaemic stroke patient 11 acute ischaemic stroke patients in the lying flat (0 degree) head position (first 24 hours of hospital admission) 11 acute ischaemic stroke patients in the sitting up ( 30 degree) head position (first 24 hours of hospital admission)
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2015-11; Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
cerebral blood flow velocity | within 24 hours, 72 hours and 3 months of the stroke symptom onset
  percentage change of the cerebral blood flow velocity in response to change of the head position within 24 hours, 72 hours and 3 months of the stroke symptom onset

SECONDARY OUTCOMES:
dynamic cerebral autoregulation | within 24 hours, 72 hours and 3 months of stroke symptom onset
  change of dynamic cerebral autoregulation within 24 hours, 72 hours and 3 months of the stroke symptom onset.
Neurovascular coupling | within 24 hours, 72 hours and 3 months of stroke symptom onset
  change of neurovascular coupling within 24 hours, 72 hours and 3 months of stroke symptom onset
Carbon dioxide reactivity | within 24 hours, 72 hours and 3 months of stroke symptom onset
  change of carbon dioxide reactivity within 24 hours, 72 hours and 3 month of stroke symptom onset.

CONTACTS AND LOCATIONS:
Overall Officials: Thompson G Robinson, MD, FRCP, Principal Investigator — University of Leicester
Locations (1):
- University Hosptial of Leicester NHS Trust, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lam MY, Haunton VJ, Nath M, Panerai RB, Robinson TG. The effect of head positioning on cerebral hemodynamics: Experiences in mild ischemic stroke. J Neurol Sci. 2020 Dec 15;419:117201. doi: 10.1016/j.jns.2020.117201. Epub 2020 Oct 21. PMID 33137635